CLINICAL TRIAL: NCT05394090
Title: The Role of Periodontal Diseases and Stimulation of Saliva Secretion in the Acute Phase of
Brief Title: The Role of Periodontal Diseases and Stimulation of Saliva Secretion in the Acute Phase of Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pomeranian Medical University
Record Dates: First submitted 2022-05-16; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Diseases; Saliva Altered; Stroke
MeSH Terms: conditions — Periodontal Diseases; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saliva-stimulated group (Experimental): In approximately 50 randomly selected patients (group 1), from the second day of admission until the end of hospitalization, a 15-minute manual stimulation of the submandibular and sublingual bib was performed internally and externally. In addition, oral hygiene was performed in patients, taking into account the tongue and cheeks.
  Interventions: Diagnostic Test: saliva stimulation
- the group in which the saliva was not stimulated (No Intervention): There was no saliva in the group of 50 patients

INTERVENTIONS:
Diagnostic Test: saliva stimulation — In 50 patients with ischemic stroke, saliva was the option of a neurologopedic massage of choice
  Arms: saliva-stimulated group

SUMMARY:
Methods: 100 consecutive patients with their first ever ischemic stroke were enrolled in the study. 56 randomly selected patients were subjected to stimulation of salivation, the remaining patients were not stimulated. The severity of the neurological condition was assessed using the NIHSS scale on days 1, 3 and 7 of stroke. The incidence of periodontal diseases was classified using the Hall's scale in the 1st day of stroke. On days 1 and 7 of stroke, the concentration of IL-1beta, MMP8, OPG and RANKL in the patients' saliva was assessed using the Elisa technique. At the same time, the level of CRP and the number of leukocytes in the peripheral blood were tested on days 1, 3 and 7 of the stroke, and the incidence of upper respiratory and urinary tract infections was assessed.

DETAILED DESCRIPTION:
The course of an ischemic stroke varies by many factors. The influence of periodontal diseases and the stimulation of salivation on the course and difficulty of stroke remains unresolved.

Methods: 100 consecutive patients with their first ever ischemic stroke were enrolled in the study. 56 randomly selected patients were subjected to stimulation of salivation, the remaining patients were not stimulated. The severity of the neurological condition was assessed using the NIHSS scale on days 1, 3 and 7 of stroke. The incidence of periodontal diseases was classified using the Hall's scale in the 1st day of stroke. On days 1 and 7 of stroke, the concentration of IL-1beta, MMP8, OPG and RANKL in the patients' saliva was assessed using the Elisa technique. At the same time, the level of CRP and the number of leukocytes in the peripheral blood were tested on days 1, 3 and 7 of the stroke, and the incidence of upper respiratory and urinary tract infections was assessed.

ELIGIBILITY:
Inclusion Criteria:

* men and women,
* at the age of 48-80,
* first-ever stroke,
* with symptoms from the anterior cerebral vascularity (basin of the internal carotid artery),
* with a significant neurological deficit (minimum 3 points according to the NIH scale)
* capable of giving informed consent;

Exclusion Criteria:

* aphasia, disturbance of consciousness, mental disorders - making it impossible to express informed consent
* surgery of the salivary glands - disrupting the secretion of saliva
* diseases of the salivary glands that disrupt the secretion of saliva (diabetes, Sjögren's syndrome, state after radiotherapy in the area of the salivary glands)

Ages: 48 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
evaluation of saliva parameters od day 1 | day 1 of stroke
  On the first day of admission, saliva (2 ml) is collected and the parameters are MMP8 (ng/mL), OPG ( (ng/mL) and RANKL (ng/mL)
evaluation of saliva parameters od day 1 | day 1 of stroke
  On the first day of admission, saliva (2 ml) is collected and the parameter IL-1Beta(pg/mL)
assessment of blood parameters from day 1 | day 1 of stroke
  Assessment of CRP(mg/L) in blood on the first day of hospitalization
assessment of blood parameters from day 1 | day 1 of stroke
  Assessment of WBC( G/µL)in blood on the first day of hospitalization

SECONDARY OUTCOMES:
evaluation of saliva parameters- second measurement | day 7 of stroke
  On the seventh day of admission, saliva (2 ml) is collected with the parameters MMP8MMP8 (ng/mL), OPG ( (ng/mL) and RANKL (ng/mL)
evaluation of saliva parameters- second measurement | day 7 of stroke
  On the seven day of admission, saliva (2 ml) is collected and the parameter IL-1Beta(pg/mL)
assessment of blood parameters from day 7 | day 7 of stroke
  Assessment of CRP(mg/L) in blood on the seven day of hospitalization
assessment of blood parameters from day 7 | day 7 of stroke
  Assessment of WBC( G/µL)in blood on the seven day of hospitalization

OTHER OUTCOMES:
Neurological assessment using the NIHSS scale | day 1 of stroke
  On admission, the patient's neurological status is assessed using the NIHSS scale
Neurological assessment using the NIHSS scale | day 3 of stroke
  On the third, the patient's neurological status is assessed using the NIHSS scale
Neurological assessment using the NIHSS scale | day 7 of stroke
  On the seventh day, the patient's neurological status is assessed using the NIHSS scale

CONTACTS AND LOCATIONS:
Overall Officials: Wioletta W Pawlukowska, dr hab., Study Chair — Department of Neurology, Pomeranian Medical University, Szczecin, Poland
Locations (1):
- Departmen of Neurology, Szczecin, Unii Lubelskiej, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pihlstrom BL, Michalowicz BS, Johnson NW. Periodontal diseases. Lancet. 2005 Nov 19;366(9499):1809-20. doi: 10.1016/S0140-6736(05)67728-8. PMID 16298220
- [Background] Blaizot A, Vergnes JN, Nuwwareh S, Amar J, Sixou M. Periodontal diseases and cardiovascular events: meta-analysis of observational studies. Int Dent J. 2009 Aug;59(4):197-209. PMID 19774803
- [Background] Mattila KJ, Asikainen S, Wolf J, Jousimies-Somer H, Valtonen V, Nieminen M. Age, dental infections, and coronary heart disease. J Dent Res. 2000 Feb;79(2):756-60. doi: 10.1177/00220345000790020901. PMID 10728977
- [Background] Hashemipour MA, Afshar AJ, Borna R, Seddighi B, Motamedi A. Gingivitis and periodontitis as a risk factor for stroke: A case-control study in the Iranian population. Dent Res J (Isfahan). 2013 Sep;10(5):613-9. PMID 24348618
- [Background] Grau AJ, Becher H, Ziegler CM, Lichy C, Buggle F, Kaiser C, Lutz R, Bultmann S, Preusch M, Dorfer CE. Periodontal disease as a risk factor for ischemic stroke. Stroke. 2004 Feb;35(2):496-501. doi: 10.1161/01.STR.0000110789.20526.9D. Epub 2004 Jan 5. PMID 14707235
- [Background] Pinho MM, Faria-Almeida R, Azevedo E, Manso MC, Martins L. Periodontitis and atherosclerosis: an observational study. J Periodontal Res. 2013 Aug;48(4):452-7. doi: 10.1111/jre.12026. Epub 2012 Dec 30. PMID 23278448
- [Background] Orlandi M, Suvan J, Petrie A, Donos N, Masi S, Hingorani A, Deanfield J, D'Aiuto F. Association between periodontal disease and its treatment, flow-mediated dilatation and carotid intima-media thickness: a systematic review and meta-analysis. Atherosclerosis. 2014 Sep;236(1):39-46. doi: 10.1016/j.atherosclerosis.2014.06.002. Epub 2014 Jun 17. PMID 25014033
- [Background] Carallo C, Fortunato L, de Franceschi MS, Irace C, Tripolino C, Cristofaro MG, Giudice M, Gnasso A. Periodontal disease and carotid atherosclerosis: are hemodynamic forces a link? Atherosclerosis. 2010 Nov;213(1):263-7. doi: 10.1016/j.atherosclerosis.2010.07.025. Epub 2010 Jul 29. PMID 20732683
- [Background] Paraskevas S, Huizinga JD, Loos BG. A systematic review and meta-analyses on C-reactive protein in relation to periodontitis. J Clin Periodontol. 2008 Apr;35(4):277-90. doi: 10.1111/j.1600-051X.2007.01173.x. Epub 2008 Feb 20. PMID 18294231
- [Result] Czlonkowska A, Ryglewicz D. [Epidemiology of cerebral stroke in Poland]. Neurol Neurochir Pol. 1999;32 Suppl 6:99-103. Polish. PMID 11107570
- Available data/document: Individual Participant Data Set — http://www.pum.edu.pl